CLINICAL TRIAL: NCT03535519
Title: Rheumatoid Arthritis Ultrasound Response to Methotrexate
Brief Title: Rheumatoid Arthritis Response to Methotrexate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Juan Carlos Nieto (Other)
Collaborators: Nordic Pharma SAS (Industry)
Responsible Party: Sponsor-Investigator, Juan Carlos Nieto, Principal investigator, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: Reuma-01-2017
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Methotrexate — standard of care treatment with methotrexate

SUMMARY:
Observational and prospective study of the ultrasound response to methotrexate in rheumatoid arthritis patients who started methotrexate

DETAILED DESCRIPTION:
* Rheumatoid arthritis patients with active disease who start subcutaneous methotrexate by their rheumatologist prescription methotrexate will be included.
* Patients will participate in a prospective and observational study in which the response to methotrexate will be assessed by ultrasound (US) of joints and tendons.
* The main objective of the study is the change in B mode and Doppler mode US after 24 weeks of methotrexate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Active rheumatoid arthritis fulfilling EULAR criteria.
* Prescription of methotrexate by a rheumatologist.
* Informed consent signed by the patient.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis fulfilling EULAR criteria with active disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasound response | Basal and at 6 months
  Change in B mode and Doppler mode synovitis and tenosynovitis

SECONDARY OUTCOMES:
Clinical response | Basal and 6 months
  Change in disease activity measured by DAS28, CDAI and SDAI
Functional response | Basal and 6 months
  Change in functional status measured by HAQ

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Nieto González, PhD, Principal Investigator — Hospital General Universitario Gregorio Maranon
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No